CLINICAL TRIAL: NCT00774046
Title: High-dose Cytarabine/Mitoxantrone Followed by Autotransplantation for Therapy-Related Myelodysplastic Syndrome/Therapy -Related Acute Myeloid Leukemia
Brief Title: High-dose Cytarabine/Mitoxantrone Followed by Autotransplantation for t-MDS/t-AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11884A
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-01

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia
Keywords: Therapy-related myelodysplastic syndrome/ Therapy -related Acute myeloid leukemia; Myelodysplastic syndrome; Acute myeloid leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Cytarabine; Mitoxantrone; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Induction chemotherapy followed by stem cell transplant (Experimental): Ara-C Mitoxantrone Etoposide Stem cell mobilization Autologous transplant
  Interventions: Drug: Ara-C; Drug: Mitoxantrone; Drug: Etoposide

INTERVENTIONS:
Drug: Ara-C — Induction: 3000mg/m2 IV infusion for day 1 and day 5
  Mobilization: within 2 weeks of end of induction therapy - 2000mg/m2 as 2 hour IV infusion once every 12 hours for 3 days (6 doses total)
  Other Names: Cytarabine; HiDAC
Drug: Mitoxantrone — Induction: 30mg/m2 after the end of HiDAC day 1 and day 5
Drug: Etoposide — Mobilization: 30mg/kg over 6 doses given once every 12 hours for 3 days
  Other Names: VP-16

SUMMARY:
The purpose of this study is to determine the effectiveness of a particular combination of drugs used to treat cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have received cytotoxic chemotherapy,radiation,or a drug known to affect the properties of DNA or cell growth for some condition other than acute myeloid leukemia prior to diagnosis.
* Patients must have t-MDS/t-AML
* To be eligible for allogeneic transplantation, patients must have a suitable donor who is HLA compatible.
* Patients must be over the age of 10.
* Patients must be reviewed and discussed at the Leukemia and Transplant Conferences of the Section of Hematology/Oncology.

Exclusion Criteria:

* Patients must not have any other serious medical condition(e.g.uncontrolled or severe cardiovascular disease, diabetes, pulmonary disease, or infection)
* Psychiatric condition which would prevent compliance or possibly be worsened by treatment

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2002-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Godley, M.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Screening
Arm/Group | Induction Chemotherapy Followed by Stem Cell Transplant
Started | 116
Completed | 60
Not Completed | 56
Not completed — Not eligible | 56
Period: Enrollment
Arm/Group | Induction Chemotherapy Followed by Stem Cell Transplant
Started | 60
Completed | 32
Not Completed | 28
Not completed — Desired other therapy/refused | 28
Period: Induction Therapy
Arm/Group | Induction Chemotherapy Followed by Stem Cell Transplant
Started | 32
Completed | 32
Not Completed | 0
Period: Stem Cell Mobilization
Arm/Group | Induction Chemotherapy Followed by Stem Cell Transplant
Started | 10 (For mobilization, the patient must have had a CR and not been a candidate for allogeneic transplant)
Completed | 7
Not Completed | 3
Not completed — Count too low (2), sudden death (1) | 3
Period: Autologous Transplant
Arm/Group | Induction Chemotherapy Followed by Stem Cell Transplant
Started | 4 (2 patients died in remission and 1 relapsed without having received transplant)
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients: Ara-C Mitoxantrone Etoposide
Arm/Group | All Patients
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 56 [23 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Response to Induction Chemotherapy (CR or PR)
Description: Complete remission (CR): <5% bone marrow blasts with recovery of peripheral blood counts; complete cytogenetic remission, the disappearance of any pre-existing cytogenetic abnormality Partial remission (PR): >5% bone marrow blasts, but less than the pre-treatment blast percentage within the bone marrow Resistant disease (RD): no significant cytoreduction in bone marrow leukemic cells from pre-treatment levels Not evaluable (NE): patients who died during induction chemotherapy or who withdrew from follow-up before assessment could be made
Time Frame: Day 28-40
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 32
percentage of participants | 81.2 [63.6 to 92.8]

2. Primary Outcome: Overall Survival
Time Frame: Up to 2000 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | All Patients
Number analyzed (Participants) | 32
Days | 399 [125 to 812]

3. Primary Outcome: Relapse-free Survival
Description: Relapse is defined as bone marrow blasts >5% if the patient had achieved a complete remission, or the recurrence of any clonal cytogenetic abnormality.
Time Frame: Up to 2000 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | All Patients
Number analyzed (Participants) | 32
Days | 415 [141 to NA] — Due to censoring, the 75th percentile was not reached.

4. Secondary Outcome: Feasibility of Stem Cell Collection
Description: Feasibility is the ability to cryopreserve >=2.0 x 10^6 CD34+ cells/kg
Time Frame: 1-5 days from initiation of stem cell collection
Population: Subset of patients in CR who underwent mobilization and attempted stem cell collection.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 10
percentage of participants | 70 [35 to 93]

5. Secondary Outcome: Numbers of Stem Cells Collected
Time Frame: 1-5 days from initiation of stem cell collection
Population: Subset of patients in CR who underwent mobilization and attempted stem cell collection.
Measure: Median (Full Range); unit: 10^6 CD34+ cells/kg
Arm/Group | All Patients
Number analyzed (Participants) | 10
10^6 CD34+ cells/kg | 4.50 [0 to 30.31]

6. Secondary Outcome: Overall Survival in Patients Undergoing Autologous Stem Cell Transplant
Time Frame: Up to 817 days
Population: Subset of patients undergoing autologous stem cell transplant
Measure: Median (Full Range); unit: Days
Arm/Group | All Patients
Number analyzed (Participants) | 4
Days | 294 [133 to NA] — Largest observation censored at 817 days

7. Secondary Outcome: Disease-free Survival in Patients Undergoing Autologous Stem Cell Transplant
Time Frame: Up to 883 days
Population: Subset of patients undergoing autologous stem cell transplant
Measure: Median (Full Range); unit: Days
Arm/Group | All Patients
Number analyzed (Participants) | 4
Days | 367 [95 to NA] — Largest observation censored at 883 days

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 7/32
Other Adverse Events (participants affected / at risk) | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=32)
Neutropenic fever (Infections and infestations) | 1 (1) — Grade 3
Infection with grade 4 neutrophils (Infections and infestations) | 3 (3)
Hemorrhage (General disorders) | 1 (1) — One intra cranial (grade 5)
Sudden death (General disorders) | 1 (1)
Hemorrhage (Gastrointestinal disorders) | 1 (1) — Grade 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=32)
Neutropenic fever (Infections and infestations) | 19 — Grade 3-4
Infection/sepsis (Infections and infestations) | 16 — Grade 3-4
Thrombocytopenia (Blood and lymphatic system disorders) | 8 — Grade 3-4
Left ventrcular dysfunction (Cardiac disorders) | 4 — Grade 3-4
Non-infectious diarrhea (Gastrointestinal disorders) | 8 — Grade 3-4
Anemia (General disorders) | 3 — Grade 3-4
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 10
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Hypotension (Cardiac disorders) | 4
Tachycardia (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 2
Mental status changes (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes